CLINICAL TRIAL: NCT00589563
Title: A Phase II Study of Sirolimus, Tacrolimus and Thymoglobulin, as Graft-versus-Host Prophylaxis in Patients Undergoing Unrelated Donor Hematopoietic Cell Transplantation
Brief Title: Sirolimus, Tacrolimus, and Antithymocyte Globulin in Preventing Graft-Versus-Host Disease in Patients Undergoing a Donor Stem Cell Transplant For Hematological Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 06141; P30CA033572 (NIH); CHNMC-06141; CDR0000579340 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-12-21; First posted 2008-01-09 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Infection; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Precancerous Condition; Secondary Myelofibrosis; Small Intestine Cancer
Keywords: graft versus host disease; infection; adult favorable prognosis Hodgkin lymphoma; adult unfavorable prognosis Hodgkin lymphoma; childhood favorable prognosis Hodgkin lymphoma; childhood unfavorable prognosis Hodgkin lymphoma; cutaneous B-cell non-Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage I adult Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; Burkitt lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent childhood anaplastic large cell lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent grade I lymphomatoid granulomatosis; recurrent grade II lymphomatoid granulomatosis; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; small intestine lymphoma; splenic marginal zone lymphoma; stage I adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult T-cell leukemia/lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult T-cell leukemia/lymphoma; stage III childhood anaplastic large cell lymphoma; stage III childhood lymphoblastic lymphoma; stage III childhood small noncleaved cell lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult T-cell leukemia/lymphoma; stage IV childhood anaplastic large cell lymphoma; stage IV childhood lymphoblastic lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); childhood acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; secondary acute myeloid leukemia; adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; accelerated phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; relapsing chronic myelogenous leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; childhood myelodysplastic syndromes; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL negative; chronic myelomonocytic leukemia; juvenile myelomonocytic leukemia; primary myelofibrosis; secondary myelofibrosis
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Infections; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precancerous Conditions; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Recurrence; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Burkitt Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic; Leukemia, Myelomonocytic, Juvenile; Primary Myelofibrosis | interventions — Antilymphocyte Serum; Cyclophosphamide; Etoposide; fludarabine phosphate; Melphalan; Methotrexate; Sirolimus; Tacrolimus; Hematopoietic Stem Cell Transplantation; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fludarabine/Melphalan Conditioning (Experimental): Fludarabine/Melphalan Conditioning with
  Sirolimus, Tacrolimus and rabbit anti-thymocyte globulin (+/- methotrexate) for GvHD Prophylaxis
  Interventions: Biological: anti-thymocyte globulin; Drug: fludarabine phosphate; Drug: melphalan; Drug: methotrexate; Drug: sirolimus; Drug: tacrolimus; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: hematopoietic stem cell transplantation; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: total-body irradiation
- FTBI/Cytoxan Conditioning (Experimental): FTBI/Cytoxan Conditioning with Sirolimus, Tacrolimus and rabbit anti-thymocyte globulin (+/- methotrexate) for GvHD Prophylaxis
  Interventions: Biological: anti-thymocyte globulin; Drug: cyclophosphamide; Drug: methotrexate; Drug: sirolimus; Drug: tacrolimus; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: hematopoietic stem cell transplantation; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: total-body irradiation
- FTBI/Etoposide Conditioning (Experimental): FTBI/Etoposide Conditioning with
  Sirolimus, Tacrolimus and rabbit anti-thymocyte globulin (+/- methotrexate) for GvHD Prophylaxis
  Interventions: Biological: anti-thymocyte globulin; Drug: etoposide; Drug: methotrexate; Drug: sirolimus; Drug: tacrolimus; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: hematopoietic stem cell transplantation; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: total-body irradiation

INTERVENTIONS:
Biological: anti-thymocyte globulin — 0.5 mg/kg on day -3, 1.5 mg/kg on day -2 and 2.5 mg/kg on day -1 or day 0 from stem cell transplant
Drug: cyclophosphamide — 60mg/kg on days -5 and -4 from stem cell transplant
  Arms: FTBI/Cytoxan Conditioning
Drug: etoposide — 60mg/kg on day -4 from stem cell transplant
  Arms: FTBI/Etoposide Conditioning
Drug: fludarabine phosphate — Fludarabine 25 mg/m2/d from days -9 to -5 from stem cell transplant
  Arms: Fludarabine/Melphalan Conditioning
Drug: melphalan — Melphalan 140 mg/m2 on day -4 from stem cell transplant
  Arms: Fludarabine/Melphalan Conditioning
Drug: methotrexate — For high risk HLA-mismatch transplant only: 5 mg/m2 on days +1, +3 and +6 from stem cell transplant
Drug: sirolimus — Adults: 12 mg loading dose on day -3 from stem cell transplant followed by 4 mg orally single morning daily dose.
  Pediatric Patients <40kg: 3 mg/m2 orally on day -3 from stem cell transplant followed by 1 mg/m2 orally single morning daily dose
Drug: tacrolimus — 0.02 mg/kd/d CIV beginning on day -3 from stem cell transplant
Procedure: allogeneic hematopoietic stem cell transplantation — The target peripheral blood stem cell dose will be 5-10 x 106/kg actual body weight
Procedure: hematopoietic stem cell transplantation — The target peripheral blood stem cell dose will be 5-10 x 106/kg actual body weight
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation — Fludarabine 25 mg/m2/d from days -9 to -5 from stem cell transplant, Melphalan 140 mg/m2 on day -4 from stem cell transplant
Procedure: peripheral blood stem cell transplantation — The target peripheral blood stem cell dose will be 5-10 x 106/kg actual body weight
Radiation: total-body irradiation — 1320 cGy in 11 fractions from day -8 to day -5 or day -9 to day -6 prior to stem cell transplant

SUMMARY:
RATIONALE: Giving chemotherapy and total-body irradiation before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving tacrolimus, sirolimus, antithymocyte globulin, and methotrexate before and after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well sirolimus, tacrolimus, and antithymocyte globulin work in preventing graft-versus-host disease in patients undergoing a donor stem cell transplant for hematological cancer .

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the incidence and severity of acute- and chronic-graft-versus-host disease (GVHD) after HLA-matched or -mismatched unrelated donor hematopoietic peripheral blood transplantation in patients with hematologic malignancies scheduled to receive immunosuppressive combination of sirolimus, tacrolimus, and anti-thymocyte globulin as GVHD prophylaxis.
* To determine the safety of this combination in the first six months post-transplant.

Secondary

* To determine the time-to-engraftment, non-relapse mortality rate, overall and disease-free survival, incidence of disease relapse, and incidence of opportunistic infections with this GVHD prophylaxis.

OUTLINE: Patients are stratified according to conditioning regimen (fludarabine phosphate and melphalan vs fractionated total-body irradiation [FTBI] and etoposide vs FTBI and cyclophosphamide) and degree of donor/recipient HLA mismatch (high-risk vs low-risk).

* Conditioning regimen: Patients receive 1 of 3 standard conditioning regimens beginning on day -9 or -8 and continuing to day -1 or 0.
* Peripheral blood stem cell transplantation: Patients receive HLA-matched or mismatched unrelated donor peripheral blood stem cells on day 0.
* Graft-versus-host disease prophylaxis: Patients receive tacrolimus IV continuously beginning on day -3 and then orally when tolerated, oral sirolimus on days -3 and -2, anti-thymocyte globulin IV over 4-8 hours on days -3 to 0, and methotrexate* IV on days 1, 3, and 6. Tacrolimus and sirolimus continue for 3-6 months (with taper).

NOTE: *Only patients with high-risk HLA mismatch receive treatment with methotrexate.

After completion of study therapy, patients are followed periodically for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hematological malignancy including any of the following:

  * Non-Hodgkin lymphoma (NHL) in any complete remission (CR) or partial response (PR)
  * Hodgkin lymphoma in any CR or PR
  * Acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) in any CR

    * Bone marrow blasts < 20% within 4 weeks of transplant and peripheral blood absolute blast count < 500/µL on the day of initiation of conditioning for patients with non-CR AML or ALL
  * Myelodysplastic syndromes (MDS) treated or untreated
  * Chronic myelogenous leukemia (CML) in chronic or accelerated phase
  * Multiple myeloma in any CR or PR
  * Chronic lymphocytic leukemia in CR or PR 2 or greater
  * Myelofibrosis and other myeloproliferative disorders

    * Bone marrow blasts < 20% within 4 weeks of transplant and peripheral blood absolute blast count < 500/µL on the day of initiation
* High-risk disease defined as AML or ALL > CR1, accelerated phase CML, recurrent aggressive lymphoma, or active lymphoproliferative disease at transplant
* Low-risk disease defined as AML or ALL in CR1, chronic phase CML, or low-grade lymphoproliferative disorder with controlled disease at transplant
* Must be planning to receive 1 of the following conditioning regimens at City of Hope:

  * Fludarabine phosphate and melphalan for patients with hematological malignancies and contraindications for conventional myeloablative regimens due to age, co-morbidity, or previous transplant
  * Fractionated total-body irradiation (FTBI) and etoposide for patients with AML and ALL or CML in accelerated phase
  * FTBI and cyclophosphamide for patients with NHL, AML, CML, and MDS
* Suitable unrelated donor available

  * HLA-matched or mismatched
  * Peripheral blood stem cells available
  * No bone marrow or ex vivo-engineered or processed graft (e.g., CD34-positive, T-cell depletion)
* No uncontrolled CNS disease

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 70-100% or ECOG PS 0-2
* Creatinine < 1.3 mg/dL or creatinine clearance ≥ 70 mL/min
* Ejection fraction > 45%
* Direct bilirubin < 3 times upper limit of normal (ULN)
* ALT and AST < 3 times ULN
* Forced vital capacity, FEV1, and DLCO > 45% of predicted
* Able to cooperate with oral medication intake
* No active donor or recipient serology positive for HIV
* No known contraindication to administration of sirolimus, tacrolimus, or anti-thymocyte globulin
* No active hepatitis B or C
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent participation in other clinical trials for prevention or treatment of viral, bacterial, or fungal disease allowed provided agents do not interact with agents used in the current study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryotaro Nakamura, MD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All patients were analyzed as a single population. Stratification by conditioning regimen was not done.
Period: Overall Study
Arm/Group | All Patients
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 59.5 [19 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 32
Diagnosis [Number; unit: participants] — Diagnosis at time of transplant.
  participants
    Acute Myeloid Leukemia | 14
    Myelodysplastic Syndrome | 6
    Acute Lymphoblastic Leukemia | 3
    Chronic Myeloid Leukemia | 3
    Non-Hodgkin Lymphoma | 3
    Myeloproliferative Disorder | 2
    Chronic Lymphocytic Leukemia | 1
Disease Status (American Society for Blood and Marrow Transplantation Guidelines) [Number; unit: participants] — Disease status at time of transplant.
  participants
    Standard Risk | 14
    High/Intermediate Risk | 18
Patient/Donor Cytomegalovirus (CMV) infection status [Number; unit: participants] — Patient CMV status listed first followed by Donor CMV status. Both are determined at time of transplant.
  participants
    Positive/Negative | 12
    Positive/Positive | 12
    Negative/Negative | 3
    Negative/Positive | 5
Human Leukocyte Antigen (HLA) Match Type [Number; unit: participants] — All mismatches occur at A, B, C, or DR.
  participants
    10/10 Matched | 18
    1 Mismatch | 12
    2 Mismatches | 1
    3 Mismatches | 1
Conditioning Regimen [Number; unit: participants]
  Fludarabine/Melphalan | 23
  Fractionated Total Body Irradiation/Cytoxan | 4
  Fractionated Total Body Irradiation/Etoposide | 5
Patient/donor sex match [Number; unit: participants]
  Male patient/Female donor | 3
  Others | 29

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Grade II-IV Acute Graft-Versus-Host Disease (GVHD) at Day 100
Description: Patients were evaluated for the development of acute GVHD within the first 100 days post HSCT. The cumulative incidence of grade II-IV acute GVHD was determined using competing risk analysis. Competing risks for acute GVHD were death and nonengraftment.
Time Frame: 100 Days Post Hematopoietic Stem Cell Transplant (HSCT)
Measure: Number (95% Confidence Interval); unit: Percentage of patients developing aGVHD
Arm/Group | All Patients
Number analyzed (Participants) | 32
Percentage of patients developing aGVHD | 37.3 [22.4 to 62.0]

2. Primary Outcome: Severity of Acute GVHD
Description: All patients were considered for the evaluation of the severity of acute GVHD.
Time Frame: 100 Days Post HSCT
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 32
participants
  No Acute GVHD | 9
  Yes - Grade I | 9
  Yes- Grade II | 9
  Yes- Grade III | 1
  Yes - Grade IV | 0
  No- Inevaluable (graft failures) | 4

3. Secondary Outcome: Time to Absolute Neutrophil Count Recovery (Engraftment)
Description: Absolute neutrophil count (ANC) recovery is defined as an ANC of ≥ 0.5 x 10^9/L (500/mm3) for three consecutive laboratory values obtained on different days
Time Frame: Patients were evaluated until neutrophil recovery, a median of 15 days post HSCT
Population: 28 of the 32 patients had absolute neutrophil count recovery.
Measure: Median (Full Range); unit: Days
Arm/Group | All Patients
Number analyzed (Participants) | 28
Days | 14.5 [10 to 26]

4. Secondary Outcome: Time to Platelet Count Recovery (Engraftment)
Description: Platelet recovery is defined as the first date of three consecutive laboratory values ≥ 25 x 10^9 L obtained on different days.
Time Frame: Patients were evaluated until platelet recovery, a median of 14 days
Population: 27 of the 32 patients had platelet recovery.
Measure: Median (Full Range); unit: Days
Arm/Group | All Patients
Number analyzed (Participants) | 27
Days | 14 [10 to 40]

5. Secondary Outcome: Occurence of Infections Including Cytomegalovirus and Epstein-Barr Virus Reactivation
Description: Participants were monitored throughout the trial (median of 28 months) for various infections/complications.
Time Frame: Median Follow Up: 28 months (Range: 1-49 months)
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 32
participants
  Neither CMV or EBV | 16
  CMV reactivation only | 9
  EBV only | 3
  Both CMV and EBV | 4

6. Secondary Outcome: Occurrence of Thrombotic Microangiopathy
Description: Participants were monitored throughout the trial (median of 28 months) for various infections/complications. This is the number of participants who developed TMA.
Time Frame: Median Follow Up: 28 Months (Range: 1-49 months)
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 32
participants | 7

7. Secondary Outcome: Occurence of Sinusoidal Obstructive Syndrome (SOS)
Description: Participants were monitored throughout the trial (median of 28 months) for various infections/complications. This is the number of participants who developed SOS.
Time Frame: Median Follow Up: 28 Months (Range: 1-49 Months)
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 32
participants | 1

8. Secondary Outcome: Non-relapse Mortality at 100 Days Post HSCT
Description: Patients were evaluated for non-relapse mortality (NRM) throughout the study. Non-relapse mortality was considered any death not attributable to relapse or disease progression. The cumulative incidence of NRM was determined using competing risk analysis. Competing risks for NRM were death due to disease progression, relapse and nonengraftment.
Time Frame: 100 day point estimate was provided
Measure: Number (95% Confidence Interval); unit: Percentage of patients with a NRM
Arm/Group | All Patients
Number analyzed (Participants) | 32
Percentage of patients with a NRM | 9.4 [3.2 to 27.5]

9. Secondary Outcome: Non-relapse Mortality at Two Years Post HSCT
Description: as for outcome 8
Time Frame: 2 year point estimate was provided.
Measure: Number (95% Confidence Interval); unit: Percentage of patients with a NRM
Arm/Group | All Patients
Number analyzed (Participants) | 32
Percentage of patients with a NRM | 15.6 [7.0 to 35.0]

10. Secondary Outcome: Overall Survival at Two Years Post HSCT
Description: Patients were evaluated for survival (OS) throughout the study. Kaplan Meier estiamtes were calculated for overall survival using time from HSCT to death of any cause or for surviving patients last contact date.
Time Frame: 2 year point estimate was provided.
Measure: Number (95% Confidence Interval); unit: Percentage of patients who died
Arm/Group | All Patients
Number analyzed (Participants) | 32
Percentage of patients who died | 65.6 [53.7 to 75.2]

11. Secondary Outcome: Event Free Survival at Two Years Post HSCT
Description: Patients were evaluated for event free survival (EFS) throughout the study. Events were defined as death, relapse, progression, or nonengraftment. Kaplan Meier estimates were calculated as time from HSCT to event.
Time Frame: 2 year point estimate was provided.
Measure: Number (95% Confidence Interval); unit: Percentage of patients with an event
Arm/Group | All Patients
Number analyzed (Participants) | 32
Percentage of patients with an event | 61.3 [49.9 to 70.8]

12. Primary Outcome: Cumulative Incidence of Chronic GVHD
Description: Patients were evaluated for the development of chronic GVHD from 101 days post HSCT to last contact or documented evidence of the disease. The cumulative incidence of chronic GVHD was determined using competing risk analysis. Competing risks for GVHD were death and nonengraftment.
Time Frame: 2 year point estimate was provided.
Measure: Number (95% Confidence Interval); unit: Percentage of patients developing cGVHD
Arm/Group | All Patients
Number analyzed (Participants) | 32
Percentage of patients developing cGVHD | 62.5 [47.8 to 81.7]

13. Primary Outcome: Severity of Chronic GVHD
Description: All Patients were considered for the evaluation of chronic GVHD severity.
Time Frame: Patients were evaluated until they developed chronic GVHD, a median of 130 days post HSCT
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 32
participants
  No Chronic GVHD | 4
  Yes- Limited | 4
  Yes - Extensive | 17
  No- Inevaluable (graft failure/died <day 100) | 7

14. Secondary Outcome: Incidence of Disease Relapse/Progression at 2 Years Post HSCT
Description: Patients were evaluated for relapse/progression post transplant throughout the study. The cumulative incidence of relapse/progression was determined using competing risk analysis. Competing risks for relapse were non-relapse mortality and nonengraftment.
Time Frame: 2 year point estimate was provided.
Measure: Number (95% Confidence Interval); unit: Percentage of patients who relapsed
Arm/Group | All Patients
Number analyzed (Participants) | 32
Percentage of patients who relapsed | 12.5 [5.0 to 31.3]

ADVERSE EVENTS:
Time Frame: 180 days
Groups:
- All Patients: All patients were analyzed as a single population. Stratification by conditioning regimen was not done. One patient did not have adverse event data collected.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 9/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=31)
Blood disorder (Blood and lymphatic system disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Ill-defined disorder (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Opportunistic infection (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=31)
Blood disorder (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 16 (16)
Hemoglobin decreased (Blood and lymphatic system disorders) | 31 (31)
Hemolysis (Blood and lymphatic system disorders) | 2 (2)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 3 (3)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 6 (6)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 2 (2)
Left ventricular failure (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 23 (23)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1)
Cushingoid (Endocrine disorders) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 3 (3)
Eye disorder (Eye disorders) | 4 (4)
Eye pain (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 3 (3)
Watering eyes (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 19 (19)
Abdominal pain (Gastrointestinal disorders) | 23 (23)
Anal pain (Gastrointestinal disorders) | 3 (3)
Ascites (Gastrointestinal disorders) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 29 (29)
Diarrhea associated with GVHD for BMT studies, if specified in the protocol. (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 12 (12)
Dysphagia (Gastrointestinal disorders) | 5 (5)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 22 (22)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Fecal incontinence (Gastrointestinal disorders) | 4 (4)
Flatulence (Gastrointestinal disorders) | 4 (4)
Gastritis (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 18 (18)
Nausea (Gastrointestinal disorders) | 29 (29)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 3 (3)
Proctitis (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 3 (3)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 25 (25)
Chest pain (General disorders) | 3 (3)
Chills (General disorders) | 25 (25)
Edema (General disorders) | 1 (1)
Edema limbs (General disorders) | 25 (25)
Facial pain (General disorders) | 4 (4)
Fatigue (General disorders) | 30 (30)
Fever (General disorders) | 19 (19)
Flu-like symptoms (General disorders) | 1 (1)
Gait abnormal (General disorders) | 2 (2)
General symptom (General disorders) | 3 (3)
Ill-defined disorder (General disorders) | 4 (4)
Injection site reaction (General disorders) | 11 (11)
Irritability (General disorders) | 1 (1)
Localized edema (General disorders) | 8 (8)
Pain (General disorders) | 17 (17)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 3 (3)
Bladder infection (Infections and infestations) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 4 (4)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 8 (8)
Infectious colitis (Infections and infestations) | 2 (2)
Lip infection (Infections and infestations) | 1 (1)
Opportunistic infection (Infections and infestations) | 11 (11)
Pancreas infection (Infections and infestations) | 2 (2)
Paranasal sinus infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6)
Sepsis (Infections and infestations) | 15 (15)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 14 (14)
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 (2)
Intraoperative venous injury - Vein-portal vein (Injury, poisoning and procedural complications) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 29 (29)
Alkaline phosphatase increased (Investigations) | 23 (23)
Amylase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 30 (30)
Bilirubin increased (Investigations) | 7 (7)
Creatine phosphokinase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 21 (21)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 4 (4)
Leukocyte count decreased (Investigations) | 31 (31)
Lipase increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 26 (26)
Neutrophil count decreased (Investigations) | 31 (31)
Neutrophils/granulocytes (ANC/AGC) for BMT studies, if specified in the protocol. (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 31 (31)
Serum cholesterol increased (Investigations) | 20 (20)
Weight gain (Investigations) | 11 (11)
Weight loss (Investigations) | 17 (17)
Acidosis (Metabolism and nutrition disorders) | 4 (4)
Alkalosis (Metabolism and nutrition disorders) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 26 (26)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 20 (20)
Blood glucose increased (Metabolism and nutrition disorders) | 31 (31)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Iron overload (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 30 (30)
Serum calcium decreased (Metabolism and nutrition disorders) | 31 (31)
Serum calcium increased (Metabolism and nutrition disorders) | 7 (7)
Serum glucose decreased (Metabolism and nutrition disorders) | 3 (3)
Serum magnesium decreased (Metabolism and nutrition disorders) | 31 (31)
Serum magnesium increased (Metabolism and nutrition disorders) | 6 (6)
Serum phosphate decreased (Metabolism and nutrition disorders) | 28 (28)
Serum potassium decreased (Metabolism and nutrition disorders) | 29 (29)
Serum potassium increased (Metabolism and nutrition disorders) | 6 (6)
Serum sodium decreased (Metabolism and nutrition disorders) | 31 (31)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 28 (28)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (16)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Buttock pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 11 (11)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 20 (20)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 6 (6)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 9 (9)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 (19)
Depressed level of consciousness (Nervous system disorders) | 5 (5)
Dizziness (Nervous system disorders) | 16 (16)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 27 (27)
Memory impairment (Nervous system disorders) | 4 (4)
Neuralgia (Nervous system disorders) | 2 (2)
Neurological disorder NOS (Nervous system disorders) | 2 (2)
Nystagmus (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (10)
Sinus pain (Nervous system disorders) | 2 (2)
Taste alteration (Nervous system disorders) | 6 (6)
Tremor (Nervous system disorders) | 9 (9)
Agitation (Psychiatric disorders) | 7 (7)
Anxiety (Psychiatric disorders) | 25 (25)
Confusion (Psychiatric disorders) | 6 (6)
Depression (Psychiatric disorders) | 12 (12)
Insomnia (Psychiatric disorders) | 24 (24)
Psychosis (Psychiatric disorders) | 1 (1)
Bladder obstruction (Renal and urinary disorders) | 1 (1)
Bladder pain (Renal and urinary disorders) | 3 (3)
Bladder spasm (Renal and urinary disorders) | 3 (3)
Bladder stenosis (Renal and urinary disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 7 (7)
Protein urine positive (Renal and urinary disorders) | 11 (11)
Renal failure (Renal and urinary disorders) | 1 (1)
Urethral pain (Renal and urinary disorders) | 5 (5)
Urinary frequency (Renal and urinary disorders) | 7 (7)
Urinary incontinence (Renal and urinary disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 6 (6)
Urogenital disorder (Renal and urinary disorders) | 4 (4)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 2 (2)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (2)
Vaginal pain (Reproductive system and breast disorders) | 2 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (23)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 (19)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 18 (18)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 15 (15)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 12 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 19 (19)
Rash desquamating (Skin and subcutaneous tissue disorders) | 28 (28)
Skin disorder (Skin and subcutaneous tissue disorders) | 10 (10)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 11 (11)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 14 (14)
Hematoma (Vascular disorders) | 6 (6)
Hemorrhage (Vascular disorders) | 4 (4)
Hypertension (Vascular disorders) | 20 (20)
Hypotension (Vascular disorders) | 17 (17)
Peripheral ischemia (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes